CLINICAL TRIAL: NCT04772625
Title: Failure Analysis of Patellofemoral Arthroplasty
Status: Active, not recruiting | Type: Observational
Sponsor: Anders Odgaard (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor-Investigator, Anders Odgaard, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: PFA_Failure_06
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Patellofemoral Osteoarthritis; Arthroplasty Complications; Knee Osteoarthritis
Keywords: Patellofemoral arthroplasty; Knee revision surgery; Indication
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- PFA: The cohort consists of all patients operated with patellofemoral arthroplasty for isolated patellofemoral osteoarthritis in Denmark from Jan 1 2008 to Dec 31 2015. The number of patients is expected to be around 500. A patellofemoral arthroplasty is defined as an arthroplasty consisting of a metal trochlear component and a polyethylene patella component. The definition of isolated patellofemoral osteoarthritis in the study is pragmatic and given by the operating surgeon.
  Interventions: Device: Patellofemoral arthroplasty

INTERVENTIONS:
Device: Patellofemoral arthroplasty — Insertion of an artificial joint between the front of the femur and the back of the patella. The femoral component consists of a metal implant, and the patellar component is a polyethylene implant. The two components replace the original articular cartilage of the patellofemoral joint.
  Other Names: Artificial joint between knee cap and thigh bone

SUMMARY:
The purpose of the retrospective cohort study is 1) to determine preoperative risk factors for revision af patellofemoral arthroplasty, and 2) to provide a detailed description of indications for revision after patellofemoral arthroplasty. All patients operated with patellofemoral arthroplasty in Denmark from January 1, 2008 to December 31, 2015, will be included in the cohort.

DETAILED DESCRIPTION:
Approx. 11,000 operations with the insertion of a knee arthroplasty (knee prosthesis) are performed annually DK. The durability and quality of the treatment are assessed with prosthesis survival, that expresses the proportion of prostheses that are still functional after a given number of years (eg the 10-year prosthesis survival for all types of knee prostheses in DK is approximately 94%).

Unicompartmental implants are increasingly used, so that only the worn part of the knee is replaced. Especially for osteoarthritis between the patella and the femur, a patellofemoral prosthesis (PFA - patellofemoral alloplasty) can be inserted, which is much smaller than the traditional full prosthesis (TKA - total knee arthroplasty).

PFA operations are controversial. A recently published Danish study (double-blind RCT) comparing TKA and PFA has shown that PFA patients achieve greater satisfaction, better knee function and greater quality of life than TKA patients. A recent study has also demonstrated that the cost of a PFA procedure is less than that of a TKA. As a paradox to this clear RCT finding, all national implant registers (Sweden, England, New Zealand, Denmark, etc.) show a significantly poorer prosthesis survival for PFA compared with TKA.

It is important for the future treatment of patients with severe osteoarthritis between the patella and femur to understand the cause of the discrepancy between RCT and registry results. The discrepancy gives rise to a number of questions regarding. indications, techniques, competences, postoperative regimens etc.

The divergence between the RCT and registry studies can only be clarified by a study that 1) examines the influence of preperative factors (patient history, physical findings, radiology etc.) on outcome, and that 2) attempts a causal analysis for each reoperation. The investigators intend to do this though a cohort study including all cases of patellofemoral arthroplasty performed in Denmark from January 1, 2008 until December 31, 2015.

The purpose is to determine preoperative risk factors for revision after PFA and to provide a detailed description of indications for revision after PFA.

ELIGIBILITY:
Inclusion Criteria:

* Patellofemoral arthroplasty
* Primary procedure performed between Jan 1 2008 and Dec 31 2015
* Primary procedure performed in Denmark

Exclusion Criteria:

* Patella-nail syndrome
* Dislocating tendon following patellectomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients operated with patellofemoral arthroplasty for patellofemoral osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Implant revision and reoperation rates | 10-year
  The proportion of revised and reoperated patients

SECONDARY OUTCOMES:
The 6-year cumulative revision rate | 6 years
  The 6-year cumulative revision rate of patellofemoral arthroplasties in a target trial comparing two groups of surgeons: 1) those surgeons, who were a part of a randomised clinical trial comparing PFA and TKA, and 2) other surgeons. In addition to this, the 6-year cumulative reoperation rate (other than revision) and the 6-year cumulative mortality rate will also be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Odgaard, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Odgaard A, Madsen F, Kristensen PW, Kappel A, Fabrin J. The Mark Coventry Award: Patellofemoral Arthroplasty Results in Better Range of Movement and Early Patient-reported Outcomes Than TKA. Clin Orthop Relat Res. 2018 Jan;476(1):87-100. doi: 10.1007/s11999.0000000000000017. PMID 29529622
- [Background] Bendixen NB, Eskelund PW, Odgaard A. Failure modes of patellofemoral arthroplasty-registries vs. clinical studies: a systematic review. Acta Orthop. 2019 Oct;90(5):473-478. doi: 10.1080/17453674.2019.1634865. Epub 2019 Jul 1. PMID 31259645
- [Background] Odgaard A, Eldridge J, Madsen F. Patellofemoral Arthroplasty. JBJS Essent Surg Tech. 2019 Apr 24;9(2):e15. doi: 10.2106/JBJS.ST.18.00094. eCollection 2019 Jun 26. PMID 31579533
- [Background] Fredborg C, Odgaard A, Sorensen J. Patellofemoral arthroplasty is cheaper and more effective in the short term than total knee arthroplasty for isolated patellofemoral osteoarthritis: cost-effectiveness analysis based on a randomized trial. Bone Joint J. 2020 Apr;102-B(4):449-457. doi: 10.1302/0301-620X.102B4.BJJ-2018-1580.R3. PMID 32228074
- [Background] Odgaard A, Kappel A, Madsen F, Kristensen PW, Stephensen S, Attarzadeh AP. Patellofemoral Arthroplasty Results in Better Time-weighted Patient-reported Outcomes After 6 Years than TKA: A Randomized Controlled Trial. Clin Orthop Relat Res. 2022 Sep 1;480(9):1707-1718. doi: 10.1097/CORR.0000000000002178. Epub 2022 Mar 21. PMID 35315804
- [Background] Rasmussen LE, Hoffmann AG, Blanche P, Espersen F, Justesen TF, Rasmussen LE, Hangaard S, Christensen R, Odgaard A. Surgeon Training and Revision Rates After Patellofemoral Arthroplasty. JAMA Netw Open. 2025 Jun 2;8(6):e2517825. doi: 10.1001/jamanetworkopen.2025.17825. PMID 40577013

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/25/NCT04772625/SAP_000.pdf